CLINICAL TRIAL: NCT06898502
Title: Investigation of Conservative Treatment Preferences of Patients With Chronic Low Back and Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sema Oztürk, master's student, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: İUCOztürk001
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low-back Pain (cLBP); Chronic Neck Pain
Keywords: chronic low back pain; chronic neck pain; physiotherapy and Rehabilitation; patitent's preference
MeSH Terms: interventions — Electric Stimulation Therapy; Transcutaneous Electric Nerve Stimulation; Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrotherapy (Experimental): All 50 patients with chronic low back pain and 50 patients with chronic neck pain will receive electrotherapy treatment, which includes TENS, hot pack, and therapeutic ultrasound methods.
  Interventions: Device: Electrotherapy ( TENS, hot pack, and therapeutic ultrasound )

INTERVENTIONS:
Device: Electrotherapy ( TENS, hot pack, and therapeutic ultrasound ) — Each participant will receive electrotherapy treatment three times a week for four weeks. Each treatment session will consist of 20 minutes of TENS, 20 minutes of hot pack, and 6 minutes of ultrasound therapy. Twelve weeks after the treatment, participants will be contacted by phone and asked about their improvement using the "Global Rating of Change Scale (GRC)." Pain intensity and disability level will be reassessed through phone interviews using the "Numeric Pain Scale," the "Oswestry Disability Index" for low back pain, and the "Neck Disability Index" for neck pain at the 12th week. Thus, it will be evaluated whether there is any difference in patient satisfaction, pain intensity, and disability at the 12th week between participants who selected electrotherapy as the most effective method and those who chose other treatments.
  Other Names: Transcutaneous Electrical Nerve Stimulation; hot pack; therapeutic ultrasound; Electrotherapy

SUMMARY:
Objective: The aim of this study is to determine the preferences of individuals with chronic low back and neck pain regarding physiotherapy treatment methods and to examine the factors influencing these preferences. Additionally, the study aims to compare patient satisfaction, pain intensity, and disability levels between individuals who receive their preferred treatment and those who do not. Moreover, the relationships between patients' demographic characteristics, pain levels, pain beliefs, disability status, and depression severity with their preferred treatment methods will be investigated.

Materials and Methods: The study will include 50 patients with chronic low back and 50 patients with neck pain. In this study, four videos introducing commonly used physiotherapy and rehabilitation methods for the treatment of low back and neck pain (electrotherapy applications -TENS, ultrasound, hot pack-, manual therapy, kinesiotaping-dry needling, education, and exercise) will be prepared and shown to the participants. Pain intensity will be assessed using the "Numeric Pain Scale," pain beliefs with the "Pain Beliefs Scale," depression severity with the "Patient Health Questionnaire," and disability level with the "Oswestry Disability Index" for low back pain and the "Neck Disability Index" for neck pain. Participants will rank the treatment methods they watched and explain their reasons for preference. Each participant will receive electrotherapy treatment three times a week for four weeks. Each treatment session will consist of 20 minutes of TENS, 20 minutes of hot pack, and 6 minutes of ultrasound therapy. Twelve weeks after the treatment, participants will be contacted by phone and asked about their improvement using the "Global Rating of Change Scale (GRC)." Pain intensity and disability level will be reassessed through phone interviews using the "Numeric Pain Scale," the "Oswestry Disability Index" for low back pain, and the "Neck Disability Index" for neck pain at the 12th week. Thus, it will be evaluated whether there is any difference in patient satisfaction, pain intensity, and disability at the 12th week between participants who selected electrotherapy as the most effective method and those who chose other treatments. Statistical analysis of the data will be conducted using the SPSS program, and the analysis results will be presented with mean, standard deviation, frequency (%), number of patients (n), and confidence interval values. Treatment preferences and the factors influencing these preferences will be statistically examined, with a significance level of p<0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the Physical Therapy Clinic of Istanbul Training and Research Hospital within the last 3 months with self-reported low back or neck pain intensity of at least 3 out of 10 on the NPRS (Numeric Pain Rating Scale),
* Patients aged 18 years or older,
* Patients who volunteered to participate in the study,
* Patients who have the ability to understand the assessment scales,
* Patients who do not have any contraindications to being included in the treatment program, These patients were included in the study.

Exclusion Criteria:

* Having undergone a physiotherapy program for low back or neck pain within the last 3 months,
* Having pain persisting for less than 3 months,
* Presence of radiculopathy or nerve root compression findings, inflammatory disease, serious metabolic, endocrine, cardiovascular, pulmonary, genitourinary, gastrointestinal, progressive/non-progressive central or peripheral neurological disease, or a history of malignancy,
* Pregnant or breastfeeding individuals, and those with serious musculoskeletal disorders other than low back or neck pain,
* Patients whose self-reported low back or neck pain intensity in the last 3 months was less than 3 out of 10 on the NPRS (Numeric Pain Rating Scale) were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | The pain intensity of all participants will be assessed using the Numeric Pain Scale (NPS) before starting the treatment and 12 weeks after the treatment.
  Patients' pain intensity will be assessed using the 10 cm Numeric Pain Scale (NPS), ranging from "0" (no pain) to "10" (unbearable pain). Patients will be asked the question, "How would you rate your current pain?" and will be requested to rate their pain on the scale.
Disability | The disability level will be assessed using the Oswestry Disability Index for low back pain and the Neck Disability Index for neck pain before starting the treatment and 12 weeks after the treatment.
  The functional disability level of patients will be determined using the Oswestry Disability Index, which evaluates daily living activities from 10 different aspects. A higher score indicates greater functional disability. The impact of neck pain on an individual's daily life will be assessed using the Neck Disability Index (NDI). The NDI consists of 10 sections that assess neck pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreational activities.
Determination of patients' treatment preferences | Patients' treatment preferences will be assessed before starting the treatment.
  In this study, To evaluate participants' perceptions regarding treatment preferences, four informative videos introducing commonly used physiotherapy and rehabilitation methods for the treatment of low back and neck pain (electrotherapy applications [TENS, ultrasound, hot pack], manual therapy, kinesiotaping and dry needling, exercise and education) will be prepared and shown to the participants. After watching the videos, participants will be asked to rank the treatment methods from the most effective to the least effective based on their perceived effectiveness, using a scale from 1 to 4 (1 = most effective, 4 = least effective).
  This ranking will be based on participants' personal evaluations and will be conducted without the use of any standardized psychometric scale. In addition, participants will be asked to explain the reasons for their preferences through open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: sema öztürk, Master's student, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Istanbul, Turkey (Türkiye)